CLINICAL TRIAL: NCT01046682
Title: Assessment of the Use of Salsalate to Decrease Endothelial Cell Activation and Inflammation in HIV-infected Adults
Brief Title: Safety and Efficacy of Salsalate to Treat Endothelial Dysfunction in HIV-infected Adults
Acronym: Salsalate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Grace McComsey, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02-08-02
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: HIV; Endothelial Dysfunction; Inflammation; Insulin Resistance
Keywords: HIV; Endothelial dysfunction; Inflammation; Insulin resistance
MeSH Terms: conditions — Inflammation; Insulin Resistance | interventions — salicylsalicylic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salsalate (Active Comparator)
  Interventions: Drug: Salsalate
- Usual care (No Intervention)

INTERVENTIONS:
Drug: Salsalate — Salsalate 2 grams orally twice a day for 13 weeks. This is the maximum dosage. During the initial 9 days of the study salsalate dose will be titrated to reach this goal dosage.
  Arms: Salsalate

SUMMARY:
This is a phase II, open label, randomized-controlled pilot study designed to study both the efficacy and safety of salsalate in decreasing endothelial cell dysfunction, systemic inflammation, and insulin resistance in HIV-infected adults. The investigators hypothesis is that salsalate will reduce inflammation and therefore endothelial cell activation and insulin resistance. The sample size will be 40, with an equal number of people being randomized to one of two groups. The first arm will be randomized to salsalate therapy. The second arm will act as a control group. The study duration will be 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. HIV-infected
3. Evidence of durable virologic suppression, i.e., must have HIV-1 RNA < 400 copies/ml at study entry and for at least 12 weeks prior to entry
4. On a stable antiretroviral (ARV) regimen, i.e., on the same ARV for at least 12 weeks prior to study entry
5. No intention to stop or modify ARV regimen during the study period

Exclusion Criteria:

1. Current pregnancy or breast feeding, or women of child bearing age who refuse or are unable to use appropriate methods for contraception during the study period
2. Any of the following conditions: diabetes (2 fasting glucose levels > 126 mg/dL or confirmed random glucose level > 200), creatinine clearance < 50, aspirin-sensitive asthma, COPD, history of bleeding gastric or duodenal ulcer, hepatic dysfunction, active hepatitis B or C, and any active infectious or inflammatory condition
3. Need for regular use of any of the following medications: salsalate, aspirin, non-steroidal antiinflammatories (NSAIDS), corticosteroids, warfarin or other anticoagulation therapy, phenytoin, valproic acid, carbonic anhydrase inhibitors, lithium, probenecid or sulfinpyrazone
4. Consumption of alcohol on a daily basis
5. Active use of illicit drugs
6. Unable to attend follow-up appointments
7. Allergy to any salicylic acid-containing medication or salsalate
8. AST or ALT > 2 upper limit of normal (ULN) within 6 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace A Mccomsey, M.D., Principal Investigator — University Hospitals Case Medical Center and Case Western Reserve University; Corrilynn O Hileman, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Hileman CO, Carman TL, Gripshover BM, O'Riordan M, Storer NJ, Harrill DE, White CA, McComsey GA. Salsalate is poorly tolerated and fails to improve endothelial function in virologically suppressed HIV-infected adults. AIDS. 2010 Jul 31;24(12):1958-61. doi: 10.1097/QAD.0b013e32833c3251. PMID 20613460

RESULTS

PARTICIPANT FLOW:
Groups:
- Salsalate: Salsalate 2 grams by mouth twice a day for a total daily dosage of 4 grams daily. Salsalate administered in 500 mg tablets. If 4 grams daily not tolerated by the participant, whatever dose up to 4 grams daily was tolerated was continues through the study.
- Usual Care: No placebo tablet was used in the study. Participants randomized to usual care received all of the study evaluations that the salsalate group did; however, no study medication was administered.
Period: Overall Study
Arm/Group | Salsalate | Usual Care
Started | 20 | 20
Completed | 18 | 20
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Salsalate | Usual Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46.5 [42.5 to 49] | 46 [44 to 52.5] | 46 [43.5 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 18 | 20 | 38
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow Mediated Dilation (FMD) of the Brachial Artery Measured by Ultrasound Over 13 Weeks
Description: Flow mediated dilation (FMD) of the brachial artery was measured by ultrasound. This is a measure of endothelial dependent endothelial cell function. Flow mediated dilation is expressed as a percent change from baseline brachial artery diameter to brachial artery diameter after reactive hyperemia. Reactive hyperemia occurred after occluding the brachial artery with a blood pressure cuff for 5 minutes.
Time Frame: Entry and week 13 visits
Population: Number of participants for analysis was determined by the number of participants that had 2 FMD tests performed
Measure: Median (Inter-Quartile Range); unit: % change from baseline
Arm/Group | Salsalate | Usual Care
Number analyzed (Participants) | 18 | 20
% change from baseline | 0.99 [-2.59 to 1.91] | -0.07 [-3.52 to 1.95]
Statistical Analysis 1: Comparison: Salsalate vs Usual Care; Using data from a different population, ie, patients with peripheral artery disease, and a different intervention, ie, omega-3 fatty acids, 15 participants were needed per group to achieve 80% power to detect a difference in means of -3.6% (the difference between the control group mean of -0.3% and a treatment group mean of 3.3%) assuming a common standard deviation of 3.3 using a two group t-test with a 0.05 two-sided significance level. 5 patients added to each arm in case nonparametric; Test type: Superiority or Other; p < 0.05, Wilcoxon rank sum test

ADVERSE EVENTS:
Arm/Group | Salsalate | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 18/20 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salsalate (N=20) | Usual Care (N=20)
Tinnitus (Ear and labyrinth disorders) | 9 (9) | 0 (0)
Transaminitis (Hepatobiliary disorders) | 8 (8) | 0 (0)
Headache (General disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Lack of placebo in the control group precluded blinding of the study investigators. Adherence was measured utilizing pill counts which assumes that pills not returned were taken by the participant. Sample size too small to detect a small effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No